CLINICAL TRIAL: NCT01593644
Title: Phase 2, Monocentric, Single Blind Study, Comparing the Efficacy and Tolerance of a Dipyridamole/Adenosine Combination Given Intravenously, as a Slow Bolus and at Low Doses to Adenosine Alone for Coronary Flow Reserve Assessment (in Patients With Stable Ischemic Heart Disease) Using Transthoracic Echodoppler
Brief Title: Phase II Study for the Diagnosis and Functional Assessment of CAD Using Transthoracic-Echodoppler
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Adenobio N.V (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: Single
Other Study IDs: ADEN-Ph2-2011-1
Record Dates: First submitted 2012-05-06; First posted 2012-05-08 (Estimated); Last update posted 2012-09-07 (Estimated); Status verified 2012-09

CONDITIONS: Ischemic Heart Disease
Keywords: Dipyridamole/adenosine combination given intravenously; slow bolus and low doses; coronary flow reserve assessment; transthoracic echodoppler; Patients; stable
MeSH Terms: conditions — Myocardial Ischemia | interventions — Adenosine; Dipyridamole; Fluid Therapy

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (1):
- adenosine + dypiridamole (Experimental)
  Interventions: Drug: adenosine + dipyridamole

INTERVENTIONS:
Drug: adenosine + dipyridamole — adenosine / dipyridamole combination given intravenously as a slow bolus at low doses
  Other Names: Adenosine : Krenosin® vials with 6 mg of adenosine in 2 ml fluid; concentration of 3 mg /ml); Dipyridamole : injectable Persantine® - vials of 10 mg/2 ml

SUMMARY:
The purpose of this study is to evaluate the efficacy and tolerance of a dipyridamole/adenosine combination given intravenously, as a slow bolus and at low doses to adenosine alone (given at its recommended dosage adjusted to patients' weight) for coronary flow reserve assessment (in 60-75 patients with stable ischemic heart disease) using transthoracic echodoppler

DETAILED DESCRIPTION:
Phase 2, monocentric, single blind study, comparing the efficacy (primary endpoint) and the safety-tolerance profile (secondary endpoint) of a dipyridamole/adenosine combination given intravenously as a slow bolus and at low doses to adenosine alone given by the same route at its standard and recommended dose.

Expected results: Non inferiority of the combination compared to standard adenosine alone in terms of hemodynamic efficacy, with maintenance of the optimal hyperemic coronary effect for at least 45 to 60 seconds after the end of the injection -Significant reduction of the incidence rate of A1 adverse events and of the severity of A2 and A1 clinical symptoms.

Primary endpoint : diastolic mean and peak coronary blood velocities Secondary endpoint : incidence rate and severity of adverse events, in particular, chest pain, dyspnoea, hypotension, bradycardia, AV blocks, arrhythmia

Number of patients: 60-75 pts with 42-50 pts acceptable for statistical analysis

Operating procedures:

Day 1 (visit): Informed consent signature, Review of inclusion and exclusion criteria, Hemodynamic variables and EKG, Cardiac history, Significant other medical diseases, Risk factors, Concomitant treatment and substances consumed within 48 hours, Transthoracic ultrasonography, Adverse events report Day 2 (telephone contact): Adverse events report

Duration of the study: 15 months

Statistical Analysis: Statistical tests will include :a paired test analysis and comparison of the means (quantitative variables) -Possibly the Mac-Nemar test for the assessment of clinical adverse events during the study test with both products.

ELIGIBILITY:
Inclusion Criteria:

* Man or post-menopausal woman or with an oral contraceptive treatment , > 18 years
* Provided written consent by patient with good understanding of the study objectives as explained by the investigator during the initial visit
* Patient with a potential or known Coronary Artery Disease
* Patient for whom transthoracic ultrasonography for coronary reserve assessment is deemed useful

Exclusion Criteria:

* Subjects under 18, pregnant or breast-feeding woman, psychotic patients or subjects placed under administrative and legal authority
* Patients judged by investigator as not able to understand the study objectives
* Patients with a medical history, in particular a heart disease history (eg AV block) judged as non eligible by investigator
* Patients whose medical treatment contra- indicates their inclusion in the study (eg chronic use of oral dipyridamole, pentoxifylline), if not stopped at least 72 hours before the study test
* Patients with symptomatic bradycardia (<40 beat/min) or with systemic hypotension (SBP > 90 mmHg
* Patients with a 2nd and 3rd degree AV block, a sick sinus syndrome, but not those with artificial pacemaker
* Patients with prolonged QT (QTc>480 ms)
* Patients with oral dipyridamole who did not stopped their medication 48hrs before the study test
* Patients who received theophylline within 5 days before study test
* Consumption of coffee, cola, tea, chocolate within 12 hrs before study test
* Patients with a history of unstable Asthma or Chronic Obstructive Pulmonary Disease with bronchoconstriction
* Patients with unstable angina pectoris or uncontrolled severe heart failure
* Patients with a recent myocardial infarction history (<7 days), or stroke episode (< 1 month)
* Patients with known TC stenosis and not yet revascularized, uncontrolled hypovolemia, known and unfixed valvular stenosis, left-right shunt, pericarditis, sympathetic nervous system dysfunction, carotid stenosis , any significant cerebrovascular insufficiency
* Patients with known allergy to adenosine or dipyridamole

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Estimated)
Dates: Start 2011-06; Primary Completion 2013-03 (Estimated)

PRIMARY OUTCOMES:
Diastolic mean and peak coronary blood velocities | 2 minutes
  hemodynamic efficacy, with maintenance of the optimal hyperemic coronary effect for at least 45 to 60 seconds after the end of the injection

SECONDARY OUTCOMES:
Incidence rate and severity of adverse events, in particular, chest pain, dyspnoea, hypotension, bradycardia, AV blocks, arrhythmia. | 24 hours
  Incidence rate of A1 adverse events and of the severity of A2 and A1 clinical symptoms

CONTACTS AND LOCATIONS:
Overall Officials: Patrick Meimoun, PhD, Principal Investigator — Centre Hospitalier de Compiègne
Locations (1):
- Centre Hospitalier de Compiègne, Compiègne, France